CLINICAL TRIAL: NCT06892951
Title: Phase I/II Safety lead-in Randomized Blind Placebo-controlled Clinical Trial: Efficacy and Safety of Caspofungin Aerosols for the Curative Treatment of Pneumocystis Pneumonia in Adjunction of Conventional Systemic Antifungal Therapy
Brief Title: CaspoNEB: Efficacy and Safety of Caspofungin Aerosols for the Curative Treatment of Pneumocystis Pneumonia
Acronym: CaspoNEB
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: University Hospital, Angers (Other Government); Centre Hospitalier Universitaire de Besancon (Other); University Hospital, Bordeaux (Other); University Hospital, Brest (Other); Centre Hospitalier Universitaire Dijon (Other); University Hospital, Grenoble (Other); University Hospital, Lille (Other); University Hospital, Limoges (Other); Hospices Civils de Lyon (Other); University Hospital, Montpellier (Other); Nantes University Hospital (Other); Centre Hospitalier Universitaire de Nice (Other); Hospital Avicenne (Other); Henri Mondor University Hospital (Other); Hopital Foch (Other); Hôpital Necker-Enfants Malades (Other); Pitié-Salpêtrière Hospital (Other); Poitiers University Hospital (Other); Reims University hospital (Other); Ohre Pharma (Unknown); Aerogen (Industry); Wako Diagnostics (Industry); Cape Cod Incorporated (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Tours university (Unknown); Amiens University Hospital (Other); Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-DR329-CaspoNEB; 2023-508861-34-00 (EU CTIS Number)
Record Dates: First submitted 2024-01-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Pneumocystis Pneumonia; Pneumocystis Jirovecii Infection; Pneumocystis Infections
Keywords: ventilation; Pneumocystis; caspofungin; echinocandin; aerosol; inhalation; nebulization; interstitial pneumonia
MeSH Terms: conditions — Pneumonia, Pneumocystis; Pneumocystis Infections; Respiratory Aspiration; Lung Diseases, Interstitial | interventions — Caspofungin

STUDY DESIGN:
Intervention Model Description: The protocol will be carried out in a sequential manner to first provide safety data and the optimal dosing regimen on inhaled caspofungin, prior to inclusion of all the other patients:
  1. Part 1: open-label, one arm, non-randomized, three centres study including six patients with ascending scheme regarding the rhythm of administration over one week, depending on the tolerance and closely monitored in intensive care unit to ensure that caspofungin is well tolerated via the inhaled route and to provide data supporting the proposed dose for part 2 (PK modeling)
  2. Part 2: comparative, two arms, add-on, multicenter, individually-randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To ensure the blind administration during the part 2, the following procedures will be carried out:
  * Central randomization by an independent statistician
  * Packaging and labelling of the intervention medications, nebulizers and tubing in such a manner that there is no way to determine to which treatment group (experimental or control) the participant is assigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 2 - randomized study (group 1) (Experimental): Conventional systemic antifungal treatment (systemic co-trimoxazole or systemic second line anti-Pneumocystis salvage therapy) + aerosols of echinocandin (50 mg caspofungin) during one to seven days (according to the regimen retained from the results of part 1 from day-1 to d-7) using vibrating mesh nebulization device
  Interventions: Drug: Caspofungin Acetate 50 MG
- Part 2 - randomized study (group 2) (Placebo Comparator): Control group: (in part 2 only) Conventional systemic antifungal treatment (systemic co-trimoxazole or systemic second-line anti-Pneumocystis salvage therapy) + aerosols of placebo (0.9% saline in a volume equivalent to the experimental group) during one to seven days (according to the regimen retained from part 1 results) using vibrating mesh nebulization device
  Interventions: Drug: Physiologic saline
- Part 1 - open study (Experimental): open-label non-randomized group, with ascending scheme regarding the dose and rhythm of administration over one week, depending on the tolerance, and closely monitored in ICU to ensure that caspofungin is well tolerated via the inhaled route, and to provide data supporting the proposed administration scheme for part 2.
  * the first two patients (included one by one) will receive two aerosols (5 mg) during the first week, four days apart on d-1 and d-5 (level 1);
  * the third and fourth will receive two aerosols (15 mg) during the first week, four days apart on d-1 and d-5 (level 2);
  * the fifth and sixth will receive two aerosols (50 mg) during the first week, four days apart on d-1 and d-5 (level 3);
  * the seventh and eighth patients will receive four aerosols (50 mg) two days apart during one week, at d-1, then d-3, d-5 and d-7 (level 4);
  * the last two patients will have daily aerosols during the first week, from d-1 to d-7 (level 5)
  Interventions: Drug: Caspofungin Acetate 50 MG

INTERVENTIONS:
Drug: Caspofungin Acetate 50 MG — The experimental treatment will be administered once daily for up to seven days, through the nebulization route by the means of a disposable vibrating mesh Aeroneb solo® nebulizer with the valved mask (Galway, Ireland). Before generating aerosol, resuspension of the caspofungin powder will be carried out in the same manner than for the IV route, into 10.5 mL saline serum. Preparation of the experimental drug (re-suspension) will be unblindly carried out in a distinct medical office by a nurse neither involved in the healthcare of the included patients, nor in the other parts of the study, data recording or outcome assessment. Once reconstituted, the suspension is expected to be limpid, with neither odour nor foam. Thereafter, its administration will be blindly completed by the clinical staff in charge of the enrolled patient.
  Arms: Part 1 - open study; Part 2 - randomized study (group 1)
Drug: Physiologic saline — Procedures will be exactly the same than those described above for the experimental group, but caspofungin will be replaced during the seven days of intervention by 10mL of 0.9% saline nebulized in the control group for a 15 minute-long process of nebulization (from d-1 to d-7).
  Arms: Part 2 - randomized study (group 2)

SUMMARY:
To assess the efficacy of administrating daily caspofungin aerosols versus placebo for seven days, in adjunction of conventional systemic antifungal therapy during curative treatment of Pneumocystis pneumonia, on the clinical outcome at the end of the nebulized therapy, in order to support a "GO / NO GO" decision towards a phase III trial of nebulized caspofungin in those patients.

DETAILED DESCRIPTION:
Pneumocystis jirovecii is an airborne-transmissible fungus which can induce pneumonia with severely impaired lung function, especially in immunocompromised patients. At least 1,000 new cases of Pneumocystis pneumonia occur each year in France with approximately 50% of cases suffering from hypoxemia. Around 15% HIV+ and 50% HIV- subjects require mechanical ventilation, and mean duration of hospitalization is about 30 days. Average mortality rate is ≈20% at 3 months, higher for critically ill patients (30%-60%).

To date, cotrimoxazole represents the gold standard anti-Pneumocystis treatment commonly associated with systemic corticosteroids in case of moderate-to-severe infection. However, treatment is long (several weeks) to achieve clearance of the fungus, which might favor lung sequelae like persistent inflammation or post-infectious fibrosis. Furthermore, therapeutic failures have been reported as high as 9-44% of patients. Five other drugs have been commonly used as curative alternatives to cotrimoxazole against P. jirovecii: pentamidine, primaquine + clindamycin, dapsone and atovaquone. Some are responsible for serious side effects, while others are complex to administer or less efficient. All exhibit clinically important drug-drug interactions. Therefore, in such a context, it is important to test new drugs and/or alternative delivery routes for existing therapies.

Echinocandin drugs, including caspofungin, are usually administered daily to treat invasive candidiasis and aspergillosis. They target the fungal cell wall, thus inhibiting the β-(1,3)-D glucan synthase enzyme. Intravenous (IV) echinocandins are generally well tolerated and are not responsibles for major drug-drug interactions. IV caspofungin was also proven effective in animal models of Pneumocystis infection and significantly improve the overall survival. Two human studies showed that in-hospital and 3-month mortality rates were similar between patients receiving daily IV echinocandin and those receiving co-trimoxazole alone. Several case reports also showed 47 successful outcomes with IV caspofungin, alone or in combination with standard treatment. A recent study reported better response and lower in-hospital mortality in patients receiving the combination of cotrimoxazole + IV caspofungin with no severe adverse events. Therefore, IV echinocandins are now recommended in the European therapeutic guidelines for non-HIV patients as a salvage therapy (CII-grade) in association with co-trimoxazole.

However, high molecular weight and elevated protein binding hamper optimal diffusion of IV caspofungin towards the lung alveoli (<5% plasma concentration), where P. jirovecii thrives. Administration through an aerosol directly delivered into the lung may circumvent this limitation. Technical feasibility of echinocandin nebulization was demonstrated in vitro with several commercial nebulizers that provided aerosol particles with adequat size and pH to ensure lung tolerance. In vivo, nebulized caspofungin, at a dosage equivalent to the usual IV dosage, showed an excellent safety profile in rats. It also reduced the fungal burden by -99% and induced elevated and prolonged concentrations of the drug in the lungs (almost 50% of the total amounts of caspofungin initially deposited into the lungs of infected rats were still detectable at 48 hours) - largely above the usual minimal inhibitory concentrations of fungal pathogens -, while caspofungin detection was almost null in other organs and blood.

Therefore, we hypothesize herein the therapeutic interest of caspofungin aerosols in adjunction with conventional antifungal therapy, as first-line curative treatment, to enhance the clinical recovery and to reduce the morbidity due to Pneumocystis pneumonia. As no clinical trials have been worldwide initiated, human efficacy and safety data of nebulized caspofungin are still lacking and will be first investigated in this study in patients. Thus organized in two successive parts, this phase I/II clinical trial represents a mandatory prelude for this original administration modality of caspofungin.

ELIGIBILITY:
Inclusion criteria:

* Male and female ≥18 years
* Medical management of Pneumocystis pneumonia based on :

  * Microbiological diagnosis of Pneumocystis pneumonia
  * Respiratory support (oxygen therapy or ventilatory assistance)
  * Systemic co-trimoxazole therapy or systemic second-line anti-Pneumocystis salvage therapy (switch to another anti-Pneumocystis drug is possible, but should be notified) (initiated within 48 hours or less before enrolment)
* Person affiliated to a French social security system or equivalent
* Written informed consent obtained from the participant or, if the patient is not able to give consent from representative (trusted person, family member) or if the delay in obtaining the consent is assumed not compatible with the enrollment requirements, a temporary approval can be obtained from the investigator. In all cases, the patient's written informed consent will have to be obtained as soon as possible.

Non-inclusion criteria:

* Persons covered by articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons: pregnant women, parturients, nursing mothers, persons deprived of their liberty by judicial or administrative decision, minors, and persons subject to a legal protection measure: guardianship or trusteeship). Pregnancy test to be performed in all women from 15 to 45 years old who have not had an ovariectomy.
* Other indication(s) for systemic administration of an echinocandin drug
* Known allergy to echinocandin drugs
* Absolute contraindication to aerosol therapy
* Concomitant co-infection at time of diagnosis (except HIV infection)
* Severe liver impairment (i.e. documented severe liver cirrhosis (Child C), or Factor-V protein < 50% and/or INR for prothrombin time of blood coagulation > 1.5)
* history of toxic epidermal necrosis (TEN) and Steven-Johnson syndrome (SJS)
* Participation in other pharmacological study that focuses on echinocandins and/or anti-infectious aerosol therapy or other anti-pneumocystis treatment
* Participation in a trial with an investigational product known to have pulmonary toxicity or of which the safety is not known

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Part 1: safety of inhaled caspofungin | D-7 (day-7)
  * frequency of adverse events
  * severity of adverse events
Part 2: proportion of patients alive and with a favorable clinical course* at the seventh day (day-7) after the first administration. | D7 (day-7)
  Composite outcome defined by at least one of the two following items persisting ≥24 hours in alive patients:
  * Relative reduction (de-escalation or withdrawal) of respiratory assistance due to clinical improvement (depending on the initial support):
    * extubation, or
    * weaning of non-invasive ventilatory support, or
    * weaning of nasal high-flow or low-flow oxygen therapy; (NB: all participating centers will implement uniform protocols for ventilatory assistance weaning)
  * Occurrence of a +50% increase in oxygenation (PaO2 / FiO2 ratio vs. the worst value observed after inclusion).

SECONDARY OUTCOMES:
Individual components of the composite primary outcome at day-7 (d-7) | D7 (day-7)
  * All-cause mortality and Pneumocystis pneumonia-related mortality
  * Improvement of respiratory function:
    * Proportion of patients alive and with relative reduction (de-escalation or withdrawal) of respiratory assistance (in percentage)
    * Proportion of patients alive and with a +50% increase in oxygenation (PaO2 / FiO2 ratio vs. the worst value observed after inclusion) (in percentage)
Safety of nebulized caspofungin in patients with Pneumocystis pneumonia through | day-1 (d-1), d-2, d-3, d-4, d-5, d-6, and d-7
  * Occurrence of serious and non-serious pulmonary adverse events and adverse effects at day-1 (d-1), d-2, d-3, d-4, d-5, d-6, and d-7 (with active monitoring of the nebulization procedure), and serious pulmonary adverse events and adverse effects at hospital discharge, d-28 and d-90
  * Occurrence of other serious adverse events and adverse effects at day-1 (d-1), d-2, d-3, d-4, d-5, d-6, d-7, hospital discharge, d-28 and d-90
  * Liver and kidney markers at day 1 (d-1), d-3, d-7, d-28 and d-90
    * transaminases (in international units/liter)
    * glutamate transferase (in international units/liter)
    * alkaline phosphatase (in international units/liter)
    * serum creatinine (in micromol/liter)
    * urea (in millimol/liter)
  * Blood counts (same dates)
    * complete blood count (in giga/liter)
    * platelets (in giga/liter)
  * Serum electrolytes (same dates)
    * sodium (in mmol/liter)
    * potassium (in mmol/liter)
    * chloride (in mmol/liter)
    * bicarbonates (in mmol/liter)
Pharmacokinetics of nebulized caspofungin | 0, 2, 4, 6, 12, 24 hours, plus residual concentration at day (d-3) and d-7
  in blood at 0, 2, 4, 6, 12, 24 hours, plus residual concentration at day-3 (d-3) and d-7 for the five first included patients receiving caspofungin, and in tracheo-bronchial aspirates at 4, 6, 24 h, at day-3 (d-3) and d-7 (or just before extubation if still alive at time of extubation) for the five first included patients receiving caspofungin and who are intubated. Caspofungin concentration measurements (in milligram/liter) will be centrally carried out at Tours university hospital at the end of the study only for patients who received nebulized caspofungin (intervention group), once the blind process will be lifted).
Mortality | day-28 (d-28) and d-90
  * All-cause at hospital discharge, day-28 (d-28) and d-90
  * Pneumocystis pneumonia-related at hospital discharge, day-28 (d-28) and d-90
Morbidity | day-1 (d-1), d-7 and d-21
  * Number of days alive without any ventilatory / oxygen support
  * Duration to clinical stability (from inclusion to hospital discharge:
    * maximum daily temperature ≤ 37.8 °C
    * maximum daily heart pace ≤ 100 bpm
    * maximum daily respiratory pace ≤ 24 cpm
    * minimum daily systolic blood pressure ≥ 90 mmHg
    * arterial oxygenation saturation ≥ 90% or PaO2 ≥ 60 mmHg while breathing room air, or PaO2/FiO2 ratio ≥ 285 mmHg, without an increase in the intensity of the ventilatory support
    * normal mental status
  * Duration of invasive ventilatory support
  * Duration of invasive and non-invasive ventilatory support
  * Duration to clinical healing :
    * clinical stability (cf. above)
    * 24h weaning of mechanical respiratory support due to patient's clinical improvement
  * Duration of hospital stay (in days)
  * Duration of ICU stay (in days)
  * Change in the sepsis-related organ failure assessments (SOFA) score
  * Requirement of a second-line (salvage) anti-Pneumocystis curative therapy (yes or no)
Pulmonary and systemic markers of lung infection (to assess the fungal clearance) | day-1 (d-1), d-3, d-7, d-28 and d-90
  * Evolution of hypoxemia:
    • alveolar-to-arterial oxygen gradient, ratio of arterial partial pressure in oxygen and pulsed oxymetry to fraction of inspired oxygen (in millimeter Hg)
  * LDH enzyme in blood (in international units/liter)
  * BDG fungal antigen in blood (in pigogram / milliliter)
  * RT-qPCR for P jirovecii nucleic acids in blood and in tracheal aspirates (in number of amplification cycles)
  * Impact on the micro-organism diversity in respiratory airways and infections
    * monitoring the expression of specific genes for distinguishing the relative representativeness between P. jirovecii asci and trophic forms from trachea-bronchial aspirates
    * identification and counting of fungal colonies from trachea-bronchial aspirates (in number of colony-forming units (CFU))
    * identification and counting of bacterial colonies from trachea-bronchial aspirates (in CFU)
  * Genotyping of P. jirovecii strains based on microsatellites markers and sequencing of DHPS/DHFR genes in respiratory fluids

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DESOUBEAUX, Prof, Study Director — University Hospital of TOURS; Stephan EHRMANN, Prof, Study Director — University Hospital of TOURS; Adrien LEMAIGNEN, Dr, Study Director — University Hospital of TOURS
Locations (1):
- CHU Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Yes
All research data can be requested
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of the study (2028)
Access Criteria: Upon request

REFERENCES:
- [Background] Limper AH. Alveolar macrophage and glycoprotein responses to Pneumocystis carinii. Semin Respir Infect. 1998 Dec;13(4):339-47. PMID 9872631
- [Background] McKinnell JA, Cannella AP, Kunz DF, Hook EW 3rd, Moser SA, Miller LG, Baddley JW, Pappas PG. Pneumocystis pneumonia in hospitalized patients: a detailed examination of symptoms, management, and outcomes in human immunodeficiency virus (HIV)-infected and HIV-uninfected persons. Transpl Infect Dis. 2012 Oct;14(5):510-8. doi: 10.1111/j.1399-3062.2012.00739.x. Epub 2012 May 1. PMID 22548840
- [Background] Lobo ML, Esteves F, de Sousa B, Cardoso F, Cushion MT, Antunes F, Matos O. Therapeutic potential of caspofungin combined with trimethoprim-sulfamethoxazole for pneumocystis pneumonia: a pilot study in mice. PLoS One. 2013 Aug 5;8(8):e70619. doi: 10.1371/journal.pone.0070619. Print 2013. PMID 23940606
- [Background] Wong-Beringer A, Lambros MP, Beringer PM, Johnson DL. Suitability of caspofungin for aerosol delivery: physicochemical profiling and nebulizer choice. Chest. 2005 Nov;128(5):3711-6. doi: 10.1378/chest.128.5.3711. PMID 16304338
- [Background] Ehrmann S, Mercier E, Vecellio L, Ternant D, Paintaud G, Dequin PF. Pharmacokinetics of high-dose nebulized amikacin in mechanically ventilated healthy subjects. Intensive Care Med. 2008 Apr;34(4):755-62. doi: 10.1007/s00134-007-0935-1. Epub 2007 Nov 29. PMID 18046534
- [Background] Beitler JR, Sarge T, Banner-Goodspeed VM, Gong MN, Cook D, Novack V, Loring SH, Talmor D; EPVent-2 Study Group. Effect of Titrating Positive End-Expiratory Pressure (PEEP) With an Esophageal Pressure-Guided Strategy vs an Empirical High PEEP-Fio2 Strategy on Death and Days Free From Mechanical Ventilation Among Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2019 Mar 5;321(9):846-857. doi: 10.1001/jama.2019.0555. PMID 30776290
- [Background] Desoubeaux G, Lemaignen A, Ehrmann S. Scientific rationale for inhaled caspofungin to treat Pneumocystis pneumonia: A therapeutic innovation likely relevant to investigate in a near future.... Int J Infect Dis. 2020 Jun;95:464-467. doi: 10.1016/j.ijid.2020.03.029. Epub 2020 Mar 16. No abstract available. PMID 32194238
- [Background] Le Gal S, Toubas D, Totet A, Dalle F, Abou Bacar A, Le Meur Y, Nevez G; Anofel Association. Pneumocystis Infection Outbreaks in Organ Transplantation Units in France: A Nation-Wide Survey. Clin Infect Dis. 2020 May 6;70(10):2216-2220. doi: 10.1093/cid/ciz901. PMID 31633150
- [Background] Desoubeaux G, Dominique M, Morio F, Thepault RA, Franck-Martel C, Tellier AC, Ferrandiere M, Hennequin C, Bernard L, Salame E, Bailly E, Chandenier J. Epidemiological Outbreaks of Pneumocystis jirovecii Pneumonia Are Not Limited to Kidney Transplant Recipients: Genotyping Confirms Common Source of Transmission in a Liver Transplantation Unit. J Clin Microbiol. 2016 May;54(5):1314-20. doi: 10.1128/JCM.00133-16. Epub 2016 Mar 2. PMID 26935726
- [Background] Alanio A, Desoubeaux G, Sarfati C, Hamane S, Bergeron A, Azoulay E, Molina JM, Derouin F, Menotti J. Real-time PCR assay-based strategy for differentiation between active Pneumocystis jirovecii pneumonia and colonization in immunocompromised patients. Clin Microbiol Infect. 2011 Oct;17(10):1531-7. doi: 10.1111/j.1469-0691.2010.03400.x. Epub 2011 Apr 12. PMID 20946413
- [Background] Nevez G, Le Gal S. Caspofungin and Pneumocystis Pneumonia: It Is Time To Go Ahead. Antimicrob Agents Chemother. 2019 Sep 23;63(10):e01296-19. doi: 10.1128/AAC.01296-19. Print 2019 Oct. No abstract available. PMID 31548210
- [Derived] Peghin M, Fishman JA, Grossi PA. Pneumocystis jiroveci: still troublesome to diagnose and treat. Curr Opin Infect Dis. 2025 Oct 18. doi: 10.1097/QCO.0000000000001155. Online ahead of print. PMID 41151592
- See also: Supplier of the device — https://www.aerogen.com/
- See also: Supplier of the drug — https://www.stragen.ch/
- See also: Supplier of the diagnostic kit — https://www.fujifilm.com/ffwk/en
- See also: Supplier of the diagnostic kit — https://www.acciusa.com/